CLINICAL TRIAL: NCT04875442
Title: Safety and Performance Study of the Electroencephalographic Recording Device and Sound Emissions MemoWave Aimed at Increasing Slow Brain Waves During Sleep to Improve Memory Consolidation in Subjects With Mild Cognitive Impairment
Brief Title: Safety and Performance Study of the Electroencephalographic Recording Device and Sound Emissions
Acronym: MEMOWAVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PROJECT STOPPED
Sponsor: BioSerenity (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2020-A01806-33
Record Dates: First submitted 2020-12-10; First posted 2021-05-06 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: The device studied is worn during the 2 polysomnogaphy nights. The device emits sounds during only one night in order to observe the difference of EEG signals.
  The night during which the device emits sounds is determined by randomization. The nature of the second night with the device, will be the reverse of the first, in a crossover fashion.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memowave emitting sound (Experimental): Patients worn Memowave during one night, and the device emits sounds to increase slow brain signals
  Interventions: Device: Memowave emitting sounds
- Memowave not emitting sound (Placebo Comparator): Patients worn Memowave during one night, and the device doesn't emit sounds
  Interventions: Device: Memowave not emitting sounds

INTERVENTIONS:
Device: Memowave emitting sounds — Memowave is worn during one night and emits sounds to increase slow brain waves
  Arms: Memowave emitting sound
Device: Memowave not emitting sounds — Memowave is worn during one night and doesn't emit sounds
  Arms: Memowave not emitting sound

SUMMARY:
Safety and performance study of the MemoWave electroencephalographic and sound recording device to increase slow brain waves during sleep to improve memory consolidation in subjects with mild cognitive impairment

DETAILED DESCRIPTION:
24 subjects aged between 40 and 85 years, presenting a mild cognitive disorder of the amnesic type (ie a memory complaint, a Mini Mental State ≥ 24 and a score ≤26 on free recall or ≤45 / 48 on total recall of the RLRI16 test) will be included;

Each patient spends 3 polysomnography nights at hospital: 1 night of habituation without Memowave device and next 2 nights with Memovave.

The device emits sounds to increase slow brain waves but Memowave emits sounds during only one of the two nights of test (night placebo vs night "verum"). The attribution of the night is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Subject presenting a mild cognitive disorder of the amnesic type, defined by a memory complaint, a Mini Mental State ≥ 24 and a score ≤26 on free recall or ≤45 / 48 on total recall) of the RLRI16 episodic verbal memory test
* At least 7 years of schooling

Exclusion Criteria:

* Severe psychiatric pathology
* Known neurological pathology
* High risk of apnea syndrome defined by at least 2 positive categories (each with a score ≥2) on the Berlin Questionnaire for Apnea Syndrome Screening
* High risk of behavioral disorder in REM sleep defined by an RBDSQ score> 5.
* Taking sleeping pills or antidepressants
* Severe heart disease or unbalanced diabetes

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
accuracy of Electroencephalography signals of Memowave | 3 days
  number of slow waves of Memomave divided by number of slow waves of Gold standard should be under 1

SECONDARY OUTCOMES:
Quality of the sleep | 3 days
  Score of 1 to 4 (where 4 is a good sleep and 1 a very bad sleep)
efficiency on mnesic consolidation | 3 days
  memory grid .More the score is high, more the efficiency is better
efficiency on mnesic consolidation | 3 days
  scale WAIS (Weschler Adult Intelligence scale). The score should be more than 100.

CONTACTS AND LOCATIONS:
Locations (1):
- ICM, Paris, France